CLINICAL TRIAL: NCT04138784
Title: Effectiveness of an Individualized Comprehensive Rehabilitation Program in Disabled Chronic Knee Osteoarthritis Women
Brief Title: Individualized Comprehensive Rehabilitation Program in Chronic Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assistant profressor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0083UG
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Rehabilitation program (Experimental): 19 women will be recruited in order to the inclusion criteria for the study and they will receive an 8-weeks individualized comprehensive rehabilitation program administered once a day.
  Interventions: Other: Individualized comprehensive rehabilitation program
- Aquatic training (Experimental): 18 women will be recruited in order to the inclusion criteria for the study and they will receive an 8-weeks hydrotherapy intervention once a day.
  Interventions: Other: Aquatic training

INTERVENTIONS:
Other: Individualized comprehensive rehabilitation program — The program general contents were pain education, joint protection techniques, general care lifestyle habits, which were complemented by a problem-based session. The program plan was designed to fit patients' goals, priorities, and lifestyles after an initial interview.
  Arms: Comprehensive Rehabilitation program
Other: Aquatic training — Patients received a 45 min-water exercise program which included balance and proprioception activities, isometric exercise, flexibility exercises, core stabilization exercises and aerobic/endurance exercises. All sessions were developed in groups and addressed by a qualified professional.
  Arms: Aquatic training

SUMMARY:
Knee osteoarthritis is a common condition characterized by pain and functional disability in older people. Prevalence increases with age and is more frequent in older women. The aim of this study was to assess the effects of an 8-weeks individualized comprehensive rehabilitation program with elastic bands on pain and functional disability in chronic knee osteoarthritis.

DETAILED DESCRIPTION:
The main symptoms of knee osteoarthritis are pain and functional disability. These symptoms are caused by a progressive loss and deterioration of articular cartilage with reactive new bone formation at the joint's surface and margins involving articular cartilage, soft tissues, and bone damage. Many treatment programs have been developed, including medication with nonsteroidal anti-inflammatory drugs, physical modalities, and therapeutic exercises. It is hypothesized that an individualized comprehensive rehabilitation program uring 8 weeks would benefit women with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary symptomatic KOA according to the criteria of the American College of Rheumatology
* Women aged older than 65 years
* Pain predominantly over the last 3 months
* Kellgren and Lawrence score ≥2.

Exclusion Criteria:

* Ankle, hip or foot severe disorders
* Chronic back pain
* Alzheimer's disease, Parkinson's disease, motor neuron disorders.
* Diabetes mellitus
* Cardiac or respiratory insufficiency
* Inability to understand the procedure

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Functionality | Baseline, 8 weeks, 3 months
  Changes in Functionality is going to be assessed by the Western Ontario and McMaster Universities (WOMAC). Scores range from 0 to 96, with higher scores indicating greater disease severity.
Changes in Physical Performance | Baseline, 8 weeks, 3 months
  Changes in Physical Performance is going to be assessed using the Stairs Climbing Test. This test assesses the ability to ascend and descend a flight of stairs, as well as lower extremity strength, power, and balance.
Changes in Physical Performance | Baseline, 8 weeks, 3 months
  Changes in Physical Performance is going to be assessed by The Timed up ad go. It involves a person standing from a 46-cm-high chair, walking 3 m, turning, walking back to the chair and sitting down.
Changes in Perceived Health Status | Baseline, 8 weeks, 3 months
  Changes in Perceived Health Status is going to be assessed by the EuroQol-5D.It contains two sections, a descriptive section and a valuation section. The descriptive section is a health status classification instrument with the following five dimensions: mobility; self-care; usual activities; pain/discomfort; and anxiety/depression. In the second section, respondents are asked to value their overall health status on a visual analogue scale ranging from 0 (defined as the worst imaginable health state) to 100 (defined as the best imaginable health state)

REFERENCES:
- [Derived] Lopez LL, Benitez PO, Lopez JC, Martos IC, Torres JR, Santiago MG, Valenza MC. Effectiveness of an individualized comprehensive rehabilitation program in women with chronic knee osteoarthritis: a randomized controlled trial. Menopause. 2022 Jun 1;29(6):687-692. doi: 10.1097/GME.0000000000001959. PMID 35674649